CLINICAL TRIAL: NCT04322266
Title: An Open-Label, Randomized, Single-Dose Crossover Study to Compare the Pharmacokinetics, Safety and Tolerability Between Fixed-Dose Combination and Co-Administration of HGP0904, HGP0608 and HCP1306 Tablets in Healthy Male Subjects
Brief Title: A Study to Compare the Pharmacokinetics, Safety and Tolerability Between Fixed-Dose Combination and Co-Administration of HGP0904, HGP0608 and HCP1306 Tablets in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-AMOS-102
Record Dates: First submitted 2019-09-09; First posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Reference-Test) (Experimental): Period1: HCP1306+HGP0904+HGP0608, Period 2: HCP1701
  Interventions: Drug: HCP1701; Drug: HCP1306; Drug: HGP0904; Drug: HGP0608
- Sequence 2 (Test-Reference) (Experimental): Period1: HCP1701, Period 2: HCP1306+HGP0904+HGP0608
  Interventions: Drug: HCP1701; Drug: HCP1306; Drug: HGP0904; Drug: HGP0608

INTERVENTIONS:
Drug: HCP1701 — Ezetimibe / Rosuvastatin / Amlodipine / Losartan potassium
Drug: HCP1306 — Ezetimibe /Rosuvastatin
Drug: HGP0904 — Amlodipine
Drug: HGP0608 — Losartan potassium

SUMMARY:
An Open-Label, Randomized, Single-Dose Crossover Study to Compare the Pharmacokinetics, Safety and Tolerability Between Fixed-Dose Combination and Co-Administration of HGP0904, HGP0608 and HCP1306 Tablets in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Age 19~45 years in healthy volunteers
2. BMI is more than 18.5 kg/m^2 , no more than 29.9 kg/m^2
3. Subjects who agree to use medically accepted dual contraceptives up to two months after the last administration date of the clinical trial drug and not to provide sperm.
4. Subjects who have ability to comprehend the objectives, contents of study and property of study drug before participating in trial and have willingness to sign of informed consent in writing

Exclusion Criteria:

1. Presence of medical history or a concurrent disease that may interfere with treatment and safety assessment or completion of this clinical study, including clinically significant disorders in digestive system, neuropsychiatric system, endocrine system, liver, cardiovascular system
2. Subjects who judged ineligible by the investigator

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2018-12-21 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Cmax of Amlodipine | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 144hours
  Pharmacokinetic evaluation
AUClast of Amlodipine | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96, 144hours
  Pharmacokinetic evaluation
Cmax of Losartan | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours
  Pharmacokinetic evaluation
AUClast of Losartan | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours
  Pharmacokinetic evaluation
Cmax of Rosuvastatin | Day 1,Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation
AUClast of Rosuvastatin | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation
Cmax of Free Ezetimibe | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation
AUClast of Free Ezetimibe | Day 1, Day15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation
Cmax of EXP3174 | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours
  Pharmacokinetic evaluation
AUClast of EXP3174 | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
Cmax of Total Ezetimibe | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation
AUClast of Total Ezetimibe | Day 1, Day 15: pre-dose(0 hour), 0.33, 0.67, 1, 1.33, 1.67, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72, 96 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Hospital (Anam), Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park JW, Chung H, Kim JM, Kim NY, Hong SH, Kim KA, Park JY. Pharmacokinetics of a Fixed-Dose Combination Product of Amlodipine, Losartan, Ezetimibe, and Rosuvastatin and Its Comparison with Co-administration of Four Individual Components in Healthy Participants. Drugs R D. 2024 Jun;24(2):179-186. doi: 10.1007/s40268-024-00460-y. Epub 2024 May 22. PMID 38775910